CLINICAL TRIAL: NCT00602082
Title: A Randomised Phase II Study Comparing Capecitabine Plus Streptozocin With or Without Cisplatin Chemotherapy as Treatment for Unresectable or Metastatic Neuroendocrine Tumors
Brief Title: Capecitabine and Streptozocin With or Without Cisplatin in Treating Patients With Unresectable or Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CRCA-CCTC-NET-01; CDR0000582315 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2004-005202-71; EU-207102; ISRCTN35124268
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-06

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Tumor
Keywords: pancreatic alpha cell adenoma; pancreatic alpha cell carcinoma; pancreatic beta islet cell adenoma; pancreatic beta islet cell carcinoma; pancreatic delta cell adenoma; pancreatic delta cell carcinoma; pancreatic G-cell adenoma; pancreatic G-cell carcinoma; gastrinoma; insulinoma; glucagonoma; pancreatic polypeptide tumor; somatostatinoma; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; islet cell carcinoma; recurrent islet cell carcinoma
MeSH Terms: conditions — Adenoma, Islet Cell; Gastrinoma; Insulinoma; Glucagonoma; Somatostatinoma; Carcinoma, Islet Cell | interventions — Capecitabine; Cisplatin; Streptozocin

INTERVENTIONS:
Drug: capecitabine
Drug: cisplatin
Drug: streptozocin
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: protein analysis
Genetic: proteomic profiling
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, streptozocin, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving capecitabine together with streptozocin is more effective with or without cisplatin in treating neuroendocrine tumors.

PURPOSE: This randomized phase II trial is studying giving capecitabine together with streptozocin to see how well it works compared with or without cisplatin in treating patients with unresectable or metastatic neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the objective response rate in patients with neuroendocrine tumors treated with capecitabine and streptozocin with or without cisplatin.

Secondary

* To determine the overall response rate, including both objective and biochemical responses, to these regimens.
* To determine the functional response to these regimens.
* To determine the toxicity of these regimens.
* To identify the optimal drug doses in each regimen to be recommended for a subsequent phase III trial.
* To determine the progression-free and overall survival of patients receiving these regimens.
* To determine the quality of life of these patients.
* To determine molecular markers predictive of response to chemotherapy.

OUTLINE: This is a multicenter study. Patients are stratified according to site of origin (known vs unknown primary site), prior antitumor treatment, tumor function (functional vs nonfunctional), and study center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive streptozocin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-21.
* Arm II: Patients receive cisplatin IV over 2 hours on day 1 and streptozocin and capecitabine as in arm I.

In both treatment arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete the EORTC QLQC30 questionnaire and EORTC QLQ-GI.NET21 module for quality-of-life assessment at baseline, every 9 weeks during treatment, and at 12 weeks post-treatment.

Tumor tissue is obtained at baseline and assessed for Ki67 and mitotic index. Novel tissue-specific transcription factors (e.g., CDX2) are also assessed. Blood samples are collected at baseline and 9 weeks and examined by DNA, RNA, and proteomic analysis.

After completion of study therapy, patients are followed every 12 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable, advanced, and/or metastatic disease meeting one of the following types:

  * Gastroentero-neuroendocrine tumor of the foregut
  * Pancreatic neuroendocrine tumor
  * Neuroendocrine tumor of unknown primary
* Measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (the longest diameter) ≥ 20 mm by conventional CT scanning or ≥ 10 mm by spiral CT scan or MRI
* No bronchial neuroendocrine tumors (NETs) or other NETs where the primary site is situated in organs above the diaphragm (e.g., laryngeal and pharyngeal NETs)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 100,000/mm³
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* AST and ALT ≤ 5 times ULN
* GFR ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No other serious or uncontrolled illness that would preclude study participation
* No medical or psychiatric condition that would influence the ability to provide consent

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior interferon therapy
* No prior systemic chemotherapy or chemotherapy administered as part of a chemo-embolization regimen, or for this condition
* No receptor-targeted radiolabeled therapy within the past 6 months
* No investigational agent within the past 4 weeks
* Prior and concurrent somatostatin analogues allowed provided symptoms are no longer controlled by this treatment or there is documented measurable disease progression on serial CT scans performed up to 6 months apart
* No palliative radiotherapy involving lesions used to measure disease

  * Palliative radiotherapy to regions not involved in measurement of disease allowed
* No other concurrent chemotherapy for this condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate

SECONDARY OUTCOMES:
Overall response rate
Functional response
Toxicity
Progression-free survival
Overall survival
Molecular markers predictive of response to chemotherapy
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Corrie, PhD, FRCP — Cambridge University Hospitals NHS Foundation Trust; Tim Meyer, MD, BSc, MRCP, PhD — University College London (UCL) Cancer Institute
Locations (17):
- United Kingdom (17):
  - Basildon University Hospital, Basildon, England
  - Addenbrooke's Hospital, Cambridge, England
  - Cookridge Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Aintree University Hospital, Liverpool, England
  - UCL Cancer Institute, London, England
  - St. Thomas' Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Royal Marsden - Surrey, Sutton, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales